CLINICAL TRIAL: NCT00789256
Title: A Pilot Study of Low Dose Melphalan and Bortezomib for Treatment of Acute Myelogenous Leukemia and High-Risk Myelodysplastic Syndromes
Brief Title: Low Dose Melphalan and Bortezomib for AML and High-Risk MDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Marc Gautier, Associate Director, Regional Affairs at Norris Cotton Cancer Center, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0337
Record Dates: First submitted 2008-10-06; First posted 2008-11-11 (Estimated); Results first posted 2013-07-22 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndromes
Keywords: Acute Myelogenous Leukemia; AML; Myelodysplastic Syndromes; MDS; Melphalan; Bortezomib; Velcade
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Melphalan; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study treatment (Experimental): All patients will receive the following regimen: 1) Melphalan 2 mg orally, once daily. 2) Bortezomib 1.0 mg/M2 IV on days 1, 4, 8, 11.
  Interventions: Drug: Melphalan; Drug: Bortezomib; Drug: Melphalan and bortezomib

INTERVENTIONS:
Drug: Melphalan — Melphalan: 2mg orally, once daily
  Other Names: Velcade
Drug: Bortezomib — Bortezomib: 1.0mg/M2 IV on days 1, 4, 8, 11
Drug: Melphalan and bortezomib

SUMMARY:
The purpose of this study is to determine the response rate of the combination of bortezomib and melphalan in patients with Acute Myelogenous Leukemia (AML) or high-risk Myelodysplastic Syndromes (MDS).

DETAILED DESCRIPTION:
In patients who develop acute myelogenous leukemia (AML) or a high-risk myelodysplastic syndrome (MDS), the current standard treatment involves multidrug induction chemotherapy utilizing an anthracycline or anthraquinone with cytarabine. While chemotherapy has proven effective at inducing remission in up to 90% of patients, elderly patients fair far worse. In patients over the age of sixty, the disease is not only less responsive to therapy, but an increased number of comorbid conditions makes induction therapy a more dangerous endeavor. Because of this, many patients are not offered standard induction chemotherapy and there is a dearth of viable alternatives for treatment of these otherwise fatal diseases.

Low dose melphalan has previously been shown to be an effective palliative treatment for patients diagnosed with AML and high-risk MDS. It was found to have an overall response rate of 40% in AML patients (30% complete remission and 10% partial remission) and a 57% overall response in high-risk MDS patients (33% complete remission, 5% partial remission, and 19% minor responses). This therapy, while not curative, is one of the few options for patients unable to tolerate more intensive treatment regimens, but desiring a potentially effective palliative regimen.

Bortezomib (VELCADE®) is an intravenously administered reversible, selective inhibitor of the 26S proteosome. Although all of the mechanisms by which this novel drug acts as an antineoplastic agent are not fully understood, in vivo and in vitro studies indicate they ultimately result in the inhibition of the gene expression necessary for cell growth and survival pathways, apoptotic pathways, and cellular adhesion, migration, and angiogenesis mechanisms.

Preclinical and clinical evaluation of the combination of melphalan and bortezomib has demonstrated impressive synergy in refractory multiple myeloma cell lines and patients with myeloma. This study aims to determine if these findings hold true in AML and MDS patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of AML or high-risk MDS Patients with chronic myelomonocytic leukemia or a refractory cytopenia with multilineage dysplasia are eligible if that have one of the following criteria:

  * >4 units of red blood cells transfused during the previous 3 months
  * platelet count <50,000/uL
  * absolute neutrophil count <1000/uL and a recent infection requiring antibiotics
* Patients may either be considered to be poor candidates for standard induction chemotherapy based on reasonable medical evidence or have declined such therapy, but still desire palliative treatment beyond that of best supportive care
* Primary refractory disease or have disease that has relapsed after prior cytoxic therapy
* Karnofsky performance status of >50%
* Patients may receive prior growth factor therapy
* Patients who received prior therapies (ex. melphalan, 5-azacitidine, low-dose cytarabine) to control their MDS or AML prior to registration (Stratum 2), but are clearly nonresponders are eligible for enrollment if expected toxicity of the prior therapy has resolved
* Voluntary written informed consent
* If female, the subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* If male, the subject agrees to use an acceptable method for contraception for the duration of the study
* Patients that have been previously treated will be eligible for study if:

  1. the previous therapy was ineffective and
  2. all expected toxicity of the previous treatment has resolved
  3. In general the following guidelines regarding the elapsed time from previous treatment to eligibility should be followed

     1. High intensity cytotoxic treatment (7&3 induction, High Dose Ara-C): 4 weeks
     2. Hematopoeitic growth factors: no delay required
     3. Low intensity treatment (such as oral melphalan or hydrea, low dose cytarabine or 5-azacitidine) No delay required if expected toxicity has resolved and regimen ineffective

Exclusion Criteria:

* AML FAB M3
* No concomitant malignancy other than a curatively treated carcinoma in situ of cervix or basal or squamous cell carcinoma of the skin
* Active, uncontrolled infections
* Chronic liver disease not due to AML, or bilirubin >2.0mg/dL
* End stage kidney disease on dialysis
* Active CNS disease. A lumbar puncture prior to treatment is not required and should not be performed in the absence of significant CNS symptoms or signs
* Patient has sensory peripheral neuropathy > grade 2 or painful peripheral neuropathy > grade 1 (see appendix A for NCI sensory neuropathy toxicity criteria) within 14 days before enrollment
* Hypersensitivity to bortezomib, boron or mannitol
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum B-human chorionic gonadotropin (B-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gautier, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Jeffrey Bubis, DO, Principal Investigator — Integrated Community Oncology Network
Locations (2):
- United States (2):
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

REFERENCES:
- [Background] Phillips GL, Reece DE, Shepherd JD, Barnett MJ, Brown RA, Frei-Lahr DA, Klingemann HG, Bolwell BJ, Spinelli JJ, Herzig RH, et al. High-dose cytarabine and daunorubicin induction and postremission chemotherapy for the treatment of acute myelogenous leukemia in adults. Blood. 1991 Apr 1;77(7):1429-35. PMID 2009367
- [Background] Johnson PR, Yin JA. Prognostic factors in elderly patients with acute myeloid leukaemia. Leuk Lymphoma. 1994 Dec;16(1-2):51-6. doi: 10.3109/10428199409114139. PMID 7696931
- [Background] Maslak PG, Weiss MA, Berman E, Yao TJ, Tyson D, Golde DW, Scheinberg DA. Granulocyte colony-stimulating factor following chemotherapy in elderly patients with newly diagnosed acute myelogenous leukemia. Leukemia. 1996 Jan;10(1):32-9. PMID 8558934
- [Background] Leith CP, Kopecky KJ, Godwin J, McConnell T, Slovak ML, Chen IM, Head DR, Appelbaum FR, Willman CL. Acute myeloid leukemia in the elderly: assessment of multidrug resistance (MDR1) and cytogenetics distinguishes biologic subgroups with remarkably distinct responses to standard chemotherapy. A Southwest Oncology Group study. Blood. 1997 May 1;89(9):3323-9. PMID 9129038
- [Background] Denzlinger C, Bowen D, Benz D, Gelly K, Brugger W, Kanz L. Low-dose melphalan induces favourable responses in elderly patients with high-risk myelodysplastic syndromes or secondary acute myeloid leukaemia. Br J Haematol. 2000 Jan;108(1):93-5. doi: 10.1046/j.1365-2141.2000.01825.x. PMID 10651730
- [Background] Omoto E, Deguchi S, Takaba S, Kojima K, Yano T, Katayama Y, Sunami K, Takeuchi M, Kimura F, Harada M, Kimura I. Low-dose melphalan for treatment of high-risk myelodysplastic syndromes. Leukemia. 1996 Apr;10(4):609-14. PMID 8618435
- [Background] Mitchell BS. The proteasome--an emerging therapeutic target in cancer. N Engl J Med. 2003 Jun 26;348(26):2597-8. doi: 10.1056/NEJMp030092. No abstract available. PMID 12826633
- [Background] King RW, Deshaies RJ, Peters JM, Kirschner MW. How proteolysis drives the cell cycle. Science. 1996 Dec 6;274(5293):1652-9. doi: 10.1126/science.274.5293.1652. PMID 8939846
- [Background] Karin M, Cao Y, Greten FR, Li ZW. NF-kappaB in cancer: from innocent bystander to major culprit. Nat Rev Cancer. 2002 Apr;2(4):301-10. doi: 10.1038/nrc780. PMID 12001991
- [Background] Haefner B. NF-kappa B: arresting a major culprit in cancer. Drug Discov Today. 2002 Jun 15;7(12):653-63. doi: 10.1016/s1359-6446(02)02309-7. PMID 12110242
- [Background] Dokter WH, Tuyt L, Sierdsema SJ, Esselink MT, Vellenga E. The spontaneous expression of interleukin-1 beta and interleukin-6 is associated with spontaneous expression of AP-1 and NF-kappa B transcription factor in acute myeloblastic leukemia cells. Leukemia. 1995 Mar;9(3):425-32. PMID 7885041
- [Background] Felix CA. Secondary leukemias induced by topoisomerase-targeted drugs. Biochim Biophys Acta. 1998 Oct 1;1400(1-3):233-55. doi: 10.1016/s0167-4781(98)00139-0. PMID 9748598
- [Background] Chernov MV, Bean LJ, Lerner N, Stark GR. Regulation of ubiquitination and degradation of p53 in unstressed cells through C-terminal phosphorylation. J Biol Chem. 2001 Aug 24;276(34):31819-24. doi: 10.1074/jbc.M103170200. Epub 2001 Jun 28. PMID 11431470
- [Background] Olsson I, Bergh G, Ehinger M, Gullberg U. Cell differentiation in acute myeloid leukemia. Eur J Haematol. 1996 Jul;57(1):1-16. doi: 10.1111/j.1600-0609.1996.tb00483.x. PMID 8698118
- [Background] Padua RA, Guinn BA, Al-Sabah AI, Smith M, Taylor C, Pettersson T, Ridge S, Carter G, White D, Oscier D, Chevret S, West R. RAS, FMS and p53 mutations and poor clinical outcome in myelodysplasias: a 10-year follow-up. Leukemia. 1998 Jun;12(6):887-92. doi: 10.1038/sj.leu.2401044. PMID 9639416
- [Background] Parry TE. The non-random distribution of point mutations in leukaemia and myelodysplasia--a possible pointer to their aetiology. Leuk Res. 1997 Jun;21(6):559-74. doi: 10.1016/s0145-2126(97)83221-3. PMID 9279367
- [Background] Rosenfeld C, Kantarjian H. Is myelodysplastic related acute myelogenous leukemia a distinct entity from de novo acute myelogenous leukemia? Potential for targeted therapies. Leuk Lymphoma. 2001 May;41(5-6):493-500. doi: 10.3109/10428190109060340. PMID 11378567
- [Background] Slingerland JM, Minden MD, Benchimol S. Mutation of the p53 gene in human acute myelogenous leukemia. Blood. 1991 Apr 1;77(7):1500-7. PMID 2009369
- [Background] Yang, H.H., et al., A phase I/II study of combination treatment with bortezomib and melphalan (Vc+M) in patients with relapsed or refractory multiple myeloma (MM). Proceedings of ASCO, 2003. Abstract 2340.
- [Background] Richardson PG, Barlogie B, Berenson J, Singhal S, Jagannath S, Irwin D, Rajkumar SV, Srkalovic G, Alsina M, Alexanian R, Siegel D, Orlowski RZ, Kuter D, Limentani SA, Lee S, Hideshima T, Esseltine DL, Kauffman M, Adams J, Schenkein DP, Anderson KC. A phase 2 study of bortezomib in relapsed, refractory myeloma. N Engl J Med. 2003 Jun 26;348(26):2609-17. doi: 10.1056/NEJMoa030288. PMID 12826635
- [Background] David P. Schenkein, M., Proteosome Inhibition, D. Jeffrey A. Bubis, Editor. 2003:Lebanon, New Hampshire.
- [Background] Cheson BD, Bennett JM, Kantarjian H, Pinto A, Schiffer CA, Nimer SD, Lowenberg B, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Wijermans PW, Gore S, Greenberg PL; World Health Organization(WHO) international working group. Report of an international working group to standardize response criteria for myelodysplastic syndromes. Blood. 2000 Dec 1;96(12):3671-4. PMID 11090046
- [Background] Common Terminology Criteria for Adverse Events. 2003, National Cancer Institute Cancer Therapy Evaluation Program.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study was open at Dartmouth-Hitchcock Medical Center, Norris Cotton Cancer Center - Manchester (NH), White River Junction Veteran's Administration Medical Center, and Integrated Community Oncology Network - Florida.
Pre-assignment Details: The intention was to accrue 13 evaluable patients for the initial stages of this study. For each strata, if there were no responders within the first 13 patients, the study would statistically rule-out a response rate of 20% or more with p = 0.05. If there were any responders, the study would accrue an additional 11 evaluable patients.
Groups:
- Strata 1: Includes patients who have not seen prior medical intervention for their disease. Patients assigned to Strata 1 will receive Melphalan 2mg orally, once daily and Bortezomib 1.0 mg/M2 IV on days 1, 4, 8, 11.
- Strata 2: Includes patients who have received prior medical intervention for their disease. Patients assigned to Strata 2 will receive Melphalan 2mg orally, once daily and Bortezomib 1.0 mg/M2 IV on days 1, 4, 8, 11.
Period: Overall Study
Arm/Group | Strata 1 | Strata 2
Started | 14 | 12
Completed | 14 (Strata 1 had 5 responders and continued accrual, but the study was closed due to low accrual.) | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Strata 1: Group 1 will include patients who have not seen prior medical intervention for their disease.
- Strata 2: will include patients who have received prior medical intervention for their disease.
- Total: Total of all reporting groups
Arm/Group | Strata 1 | Strata 2 | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 5 | 5
  >=65 years | 14 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (4.53) | 68 (9.07) | 71 (7.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of the Combination of Bortezomib and Melphalan in Patients With AML and High-risk MDS.
Description: Determine disease response to treatment using Cheson 2000 report of an international working group to standardize response criteria for myelodysplastic syndromes.
Time Frame: Post Cycle 1 through 28 days post-treatment
Measure: Number; unit: participants
Arm/Group | Strata 1 | Strata 2
Number analyzed (Participants) | 14 | 12
participants | 5 | 2

2. Secondary Outcome: Determine Safety Profile of the Combination of Bortezomib and Melphalan.
Description: The safety profile is based on the number of adverse events experienced by participants as reported in the Adverse Events results section for this protocol.
Time Frame: Start of treatment through 28 days post-treatment
Measure: Count of Participants; unit: Participants
Groups:
- Study Treatment: All patients will receive the following regimen: 1) Melphalan 2 mg orally, once daily. 2) Bortezomib 1.0 mg/M2 IV on days 1, 4, 8, 11.
  Melphalan: Melphalan: 2mg orally, once daily
  Bortezomib: Bortezomib: 1.0mg/M2 IV on days 1, 4, 8, 11
  Melphalan and bortezomib
Arm/Group | Study Treatment
Number analyzed (Participants) | 26
Participants
  Reported adverse events | 24
  Without reportable adverse event | 2

3. Secondary Outcome: Number of Participants With Correlation Between in Vitro and in Vivo Activity of the Combination of Bortezomib and Melphalan.
Description: Leukemic cells will be collected to test the presence of the study drugs using a cell viability assay in vitro and in vivo.
Time Frame: Pre-treatment and at complete response
Population: No data was collected and these results were not obtained. The collaborating laboratory with the capability to perform the assay with leukemic cells was not available to analyze the samples.
Arm/Group | Strata 1 | Strata 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Strata 1 | Strata 2
Serious Adverse Events (participants affected / at risk) | 1/14 | 3/12
Other Adverse Events (participants affected / at risk) | 14/14 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strata 1 (N=14) | Strata 2 (N=12)
Febrile neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Legionella Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
CNS Hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Strata 1 (N=14) | Strata 2 (N=12)
Neutropenia (Blood and lymphatic system disorders) | 10 (10) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (10) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Zoster reactivation (Infections and infestations) | 1 (1) | 0 (0)
Infection NOS (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Febrile neutropenia (Infections and infestations) | 3 (3) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Generalized weakness (General disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No